CLINICAL TRIAL: NCT03602287
Title: Effect of 2% Lignocaine Solution in Pain During Removal of Nasal Pack
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the article is not a clinical trial but is a hospital based randomized comparative study. This was inadvertently uploaded.
Sponsor: Dhulikhel Hospital (Other)
Responsible Party: Principal Investigator, Dr Ashish Dhakal, Lecturer, Dhulikhel Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14/18
Record Dates: First submitted 2018-07-07; First posted 2018-07-26 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Nasal Pack Removal
Keywords: anterior nasal pack; nasal pack removal; 2% lignocaine
MeSH Terms: interventions — Lidocaine; Injections; Pharmaceutical Preparations; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2% lignocaine (Active Comparator): In the Lignocaine group, 2.5 ml of 2% of lignocaine is diluted with 2.5 ml of distilled water, and the 5ml solution will be injected into the Merocel pack 15 minutes before removal of the pack. Nothing will be done to the opposite nostril, which would act as a control.
  Interventions: Drug: Lignocaine 2% Injection 20Ml Vial (Product)
- Normal saline (Placebo Comparator): In the Normal saline group, 5 ml of normal saline was injected into the Merocel pack 15 minutes before removal of the pack. Nothing will be done to the opposite nostril.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lignocaine 2% Injection 20Ml Vial (Product) — 2.5 ml of 2% of lignocaine is diluted with 2.5 ml of distilled water, and the 5ml solution will be injected into the Merocel pack 15 minutes before removal of the pack
  Arms: 2% lignocaine
Drug: Normal saline — 5 ml of normal saline was injected into the Merocel pack 15 minutes before removal of the pack
  Arms: Normal saline

SUMMARY:
To evaluate the efficacy of rehydration of Merocel nasal packs with 2% Lignocaine on reducing pain and discomfort during nasal pack removal in patients undergoing septoplasty.

DETAILED DESCRIPTION:
This study will be carried out in patients who have undergone septoplasty for deviated nasal septum under general anesthesia, and who are categorized as American Society of Anesthesiologists (ASA) grade I to II. Consent will be obtained from the patient for the same.

Septoplasty will be carried out under general anesthesia and in all patients Merocel nasal packs (expandable polyvinyl acetate nasal packing) that expand upon contact with fluid will be used.

The postoperative analgesia will include Ibuprofen 400mg + Paracetamol 500mg combination thrice daily and Ketorolac 30mg intravenous when needed. The packs will be removed on the second postoperative day, 48 hours after packing.

During nasal pack removal, the subjects will be randomly divided into 2 groups: the Lignocaine group (2% lignocaine HCl) and the Normal saline group (0.9% NaCl) using simple random sampling by lottery method. Subjects won't know which group they belong to and what medication they will be receiving. A 23-gauge needle will be used for direct application of the treatment to the Merocel, with care taken not to touch the patient.

In the Lignocaine group, 2.5 ml of 2% of lignocaine is diluted with 2.5 ml of distilled water, and the 5ml solution will be injected into the Merocel pack 15 minutes before removal of the pack. Nothing will be done to the opposite nostril, which would act as a control.

In the Normal saline group, 5 ml of normal saline was injected into the Merocel pack 15 minutes before removal of the pack. Nothing will be done to the opposite nostril.

All patients will be blinded to which group they belong and which solution was being kept in their pack.

All patients will be asked to evaluate the severity of pain during removal of nasal packing by Visual Analogue Scale (VAS) (range, 0-10; 0 = no pain and 10 = intolerable pain).

Adverse events such as vomiting and nausea will be recorded. These procedures will be done by the same team to minimize observer variations.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic deviated nasal septum undergone Septoplasty surgery with bilateral anterior nasal packing

Exclusion Criteria:

* History of previous nasal surgeries
* Nasal polyposis
* Allergic rhinitis
* Chronic sinusitis
* Patient with neurological and psychiatric disease
* Patient with sensitivity to anesthetic agent in study
* Patients unwilling to enroll in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
This study is used to determine whether re-hydrating Merocel nasal packs with 2% Lignocaine reduces pain during nasal pack removal. | During Nasal pack removal at 48 hrs post operative
  Post-operative pain severity was assessed with Visual Analogue Scale (VAS). It's a 10cm scale in which 0 represents no pain at all and 10 represents the worst pain imaginable. This would find out if rehydrating nasal pack with mentioned material decreases pain caused to the patient during pack removal.

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Dhakal, Principal Investigator — Dhulikhel Hospital
Locations (1):
- Dhulikhel Hospital, Dhulikhel, Kavre, Nepal

IPD SHARING:
Plan to Share IPD: Undecided